CLINICAL TRIAL: NCT06944717
Title: A Phase 1, Single Center, Open Label, Single Dose, Dose Escalation Study to Determine the Safety and Immunogenicity of a Novel Bivalent Norovirus G1.1 and G2.4 Vaccine Administered Orally to Healthy Volunteers Aged ≥ 18 Years and ≤ 80 Years Old
Brief Title: A Trial of a Norovirus G1.1 and G2.4 Vaccine Administered Orally to Healthy Participants Aged ≥ 18 Years and ≤ 80 Years Old
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: VXA-NVV-109
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Norovirus Infections
Keywords: Norovirus; Healthy participants; VXA-G1.1-NN; VXA-G2.4-NS; VXA-G2.4-NS-T; VXA-G1.1-NN-T
MeSH Terms: conditions — Caliciviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Bivalent Low Dose Next Generation Vaccine (Experimental): Healthy participants will receive Norovirus GI.1 Norwalk VP1 Vaccine, Modified Oral E1-/E3-Deleted Replication Defective Recombinant Adenovirus 5 with dsRNA Adjuvant (VXA-G1.1-NN-T) (1x10^10 infectious units (IU)) and Norovirus GII.4 Sydney VP1 Vaccine, Modified Oral E1-/E3-Deleted Replication Defective Recombinant Adenovirus 5 with dsRNA Adjuvant (VXA-G2.4-NS-T) (1x10^10 IU) orally.
  Interventions: Biological: VXA G1.1 NN-T; Biological: VXA G2.4 NS-T
- Bivalent High Dose Legacy Vaccine (Experimental): Healthy participants will receive Norovirus GI.1 Norwalk Vaccine Protein 1 (VP1) Vaccine, Oral E1-/E3-Deleted Replication Defective Recombinant Adenovirus 5 with double-stranded ribonucleic acid (dsRNA) Adjuvant (VXA-G1.1-NN) (1x10^11 IU) and Norovirus GII.4 Sydney VP1 Vaccine, Oral E1-/E3-Deleted Replication Defective Recombinant Adenovirus 5 with dsRNA Adjuvant (VXA-G2.4-NS) (1x10^11 IU) orally.
  Interventions: Biological: VXA-G1.1-NN; Biological: VXA-G2.4-NS
- Bivalent High Dose Next Generation Vaccine (Experimental): Healthy participants will receive VXA-G1.1-NN-T (1x10^11 IU) and VXA-G2.4-NS-T (1x10^11 IU) orally. A sentinel group will be enrolled, if there is positive recommendation from the safety monitoring committee, enrollment will continue in this arm.
  Interventions: Biological: VXA G1.1 NN-T; Biological: VXA G2.4 NS-T

INTERVENTIONS:
Biological: VXA-G1.1-NN — Legacy vaccine, administered orally.
  Arms: Bivalent High Dose Legacy Vaccine
Biological: VXA-G2.4-NS — Legacy vaccine, administered orally.
  Arms: Bivalent High Dose Legacy Vaccine
Biological: VXA G1.1 NN-T — Next generation vaccine, administered orally.
  Arms: Bivalent High Dose Next Generation Vaccine; Bivalent Low Dose Next Generation Vaccine
Biological: VXA G2.4 NS-T — Next generation vaccine, administered orally.
  Arms: Bivalent High Dose Next Generation Vaccine; Bivalent Low Dose Next Generation Vaccine

SUMMARY:
The primary objective of this study is to determine the safety and immunogenicity of low and high dose regimens of a next generation norovirus bivalent G1.1 and G2.4 vaccine candidate in healthy participants.

ELIGIBILITY:
Inclusion Criteria

1. ≥ 18 and ≤ 80 years old at the time of signing the Informed Consent Form (ICF).
2. In stable and good general health and without significant medical illness (based on review of medical history, physical examination, current health status, and vital signs at Screening) as determined by the Investigator, with Screening lab values within normal limits or abnormalities assessed as not clinically significant.
3. Body mass index (BMI) > 17.0 and < 35.0 kg/m^2 at Screening.
4. Available for all planned visits and tele-health appointments, and willing to complete all Protocol-defined procedures and assessments (including ability and willingness to swallow multiple small enteric-coated tablets per study dose).
5. Male or female participants.

   1. Female participants must not be breastfeeding and must provide a negative pregnancy test at Screening and pre-dose on Day 0.
   2. Female participants must fulfill at least one of the following criteria:

      * At least 1 year post-menopausal (defined as amenorrhea for ≥ 12 consecutive months prior to Screening without alternative medical cause) or surgically sterile (hysterectomy, bilateral salpingectomy, bilateral oophorectomy, bilateral tubal occlusion/ligation).
      * Female participants of childbearing potential must be willing to use a highly effective form of contraception for 30 days prior to study drug administration and until 60 days after study drug administration. Acceptable forms are oral, implantable, intrauterine, transdermal, intravaginal, injectable, double barrier or abstinence (participants using diaphragms must also use condoms). The Investigator must approve the form of contraception. Female participants must also refrain from egg donation for the 1 month prior to dosing through 60 days post-vaccination.
   3. Male participants must fulfill one of the following criteria:

      * Male participants must agree to refrain from donating sperm and practice abstinence from all intercourse or use an effective method of birth control which includes condom use from study drug administration to 90 days post-dose.
      * At least 1 year post-vasectomy and have confirmed that they have obtained documentation of the absence of sperm in the ejaculate.
6. Capable of understanding and giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in the Protocol.

Exclusion Criteria

1. Presence of significant uncontrolled medical or psychiatric illness (acute or chronic) including institution of new medical/surgical treatment or significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months prior to Screening and reconfirmed at baseline.
2. Cancer, or treatment for cancer or any procedure or preventive medication for cancer or to prevent recurrence, within past 3 years (excluding fully treated and resolved basal cell carcinoma or squamous cell carcinoma).
3. Presence of immunosuppression or medical condition possibly associated with impaired immune responsiveness, including diabetes mellitus- type 1 and 2, asplenia, and functional asplenia.
4. History of irritable bowel disease or other inflammatory digestive or gastrointestinal condition that could affect the distribution/safety evaluation of an orally administered vaccine targeting the mucosa of the small intestine. Such conditions may include but are not limited to:

   1. Any history of:

      * Gastrointestinal malignancy
      * Masabsorption
      * Pancreato-biliary disorders
      * Inflammatory bowel disease
      * Irritable bowel disease
      * Hiatal hernia
      * Surgical resection
   2. History of diagnosis or treatment in past 5 years of:

      * Osophageal or gastric motility disorder
      * Gastro esophageal reflux disorder if any of the following is met:

        * History of severe or uncontrolled gastroesophageal reflux disease (GERD) at any point during this period.
        * History of complicated GERD at any point during this period.
        * Was on treatment for 12 continuous weeks at any point during this period.
        * Has been with chronic or frequent GERD symptoms (e.g., more than twice per week) in the past year.
      * Peptic ulcer if any of the following is met:

        * History of severe or uncontrolled peptic ulcer at any point during this period.
        * History of complicated peptic ulcer at any point during this period.
        * Was on treatment for 12 continuous weeks at any point during this period.
        * Has been with chronic or frequent peptic ulcer symptoms (e.g., more than twice per week) in the past year.
      * Cholecystectomy if any of the following is met:

        * Procedure was performed within 1 year of dosing.
        * The participants has ongoing / unresolved post-cholecystectomy digestive symptoms within 30 days prior to dosing.
5. History of any form of angioedema.
6. History of serious reactions to vaccination such as anaphylaxis, respiratory problems, hives, or abdominal pain.
7. Known contraindication to blood draws (e.g., bleeding diathesis, acquired coagulopathy, significant bleeding, or bruising) or to oral route of administration (unable to swallow tablets).
8. Has an acute disease within 72 hours prior to study drug administration, defined as the presence of a moderate or severe illness (as determined by the Investigator through medical history and physical exam), including the following (Note: Assessment may be repeated once during Screening Period):

   1. An acute illness that is nearly resolved, with only minor residual symptoms remaining, is allowable if, in the opinion of the site investigator, the residual symptoms will not interfere with the ability of study staff to assess safety parameters as required by the Protocol.
   2. Presence of a fever ≥ 38.0°C (100.4°F) measured orally at baseline on Day 1 prior to dosing.
   3. Receipt of antipyretic/analgesic medications within 24 hours prior to vaccine administration.
9. Any significant hospitalization within the last year which in the opinion of the Investigator or Sponsor could interfere with study participation.
10. Any of the following personal and/or family history or conditions that may lead to higher risk of clotting events and/or thrombocytopenia:

    1. Familial coagulopathy or hypercoagulability or personal history of bleeding disorder or thrombosis/embolus.
    2. History of heparin-related thrombotic events, and/or receiving heparin treatments.
    3. History of autoimmune or inflammatory disease such as autoimmune thyroiditis, vitiligo, rheumatoid arthritis.
    4. Presence of any of the following conditions known to increase risk of thrombosis within 6 months prior to Screening:

       * Recent surgery other than removal/biopsy of cutaneous lesions.
       * Immobility (confined to bed or wheelchair for 3 or more successive days).
       * Head trauma with loss of consciousness or documented brain injury.
       * Receipt of anticoagulants for prophylaxis of thrombosis.
       * Recent clinically significant infection, including hospitalization for Coronavirus Disease 19 (COVID-19) related illness.
11. Any other condition that in the clinical judgement of the investigator would jeopardize the safety or rights of a participant taking the study drug, would render the participant unable to comply within the Protocol or would interfere with the evaluation of the study endpoints diagnostic assessments including a history of drug, alcohol, or chemical abuse within 1 year of Screening.
12. Positive human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) tests at the Screening visit.
13. History of gastrointestinal bleeding including hematochezia (blood in stool) or melena (black stool) of unknown etiology or that has not been evaluated.
14. Positive urine drug screen (UDS) for drugs of abuse at Screening (positive test for marijuana is not exclusionary; however concurrent use of marijuana during the Active Study Period through Day 28 is prohibited). Positive UDS at Screening due to prescribed stimulants will be reviewed on a case by case basis.
15. Positive breath or urine alcohol test at baseline (prior to dosing).
16. Receipt of a licensed vaccine (including any COVID-19 vaccines under Emergency Use Authorization [EUA]) within 14 days prior to study drug administration or planned administration during the Active Study Period (Day 28).
17. Use of antibiotics, proton pump inhibitors, H2 blockers or antacids within 7 days prior to study drug administration or planned use during the active study period (up to Day 28).
18. Use of drugs known to affect gastrointestinal motility including glucagon-like peptide 1 receptor agonists including tirzepatide (Mounjaro) and semaglutide (Wegovy, Ozempic) within 30 days prior to drug administration or planned use through Day 7. Okay to restart after Day 7 if with full resolution of solicited symptoms of reactogenicity.
19. Use of medications known to affect the immune function (e.g., including but not limited to corticosteroids (systemic, intranasal, inhaled, or intra-articular), leukotriene modifiers, and Janus kinase inhibitors) within 14 days before study drug administration or planned use during the Active Study Period (up to Day 28).

    a. Exception to the timeframe: allergen immunotherapy (AIT) will be allowed only if the participant is stable in the maintenance phase of AIT. Maintenance AIT should not be dosed for at least 7 days before and 7 days after study vaccine dosing, and the Principal Investigator must document the treating allergist's approval.
20. Daily use of nonsteroidal anti-inflammatory drugs within 7 days prior to study drug administration or planned use during the active study period (up to Day 28). Low daily doses of acetylsalicylic acid ≤ 100 mg for cardio-protection is not exclusionary.
21. Administration of any investigational vaccine, drug or device within 8 weeks preceding study drug administration, or planned use within the duration of the study.
22. Previous participation in a Vaxart Clinical Trial or other norovirus vaccine trial unless confirmed receipt of placebo.
23. Donation or use of blood or blood products within 30 days prior to study drug administration or planned donation during the active study period (up to Day 28).
24. History of hypersensitivity or allergic reaction to any component of the investigational vaccine, including but not limited to, fish gelatin allergy.
25. Study team member or first-degree relative of any study team member (inclusive of Sponsor and site personnel involved in the study).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Solicited Symptoms of Reactogenicity (Gastrointestinal and Systemic) for 1 Week Following Study Intervention Dose | 7 days
Duration of Solicited Symptoms of Reactogenicity (Gastrointestinal and Systemic) for 1 Week Following Study Intervention Dose | Approximately 1 year
Severity of Solicited Symptoms of Reactogenicity (Gastrointestinal and Systemic) for 1 Week Following Study Intervention Dose | 7 days
Number of Participants Experiencing Unsolicited Adverse Events (AE) for 28 Days Following the Study Intervention Dose | 28 days
Number of Participants Experiencing Unsolicited New Onset of Chronic Illness (NOCI) for 28 Days Following the Study Intervention Dose | 28 days
Duration of Unsolicited AEs for 28 Days Following the Study Intervention Dose | Approximately 1 year
Duration of Unsolicited NOCIs for 28 Days Following the Study Intervention Dose | Approximately 1 year
Severity of Unsolicited AEs for 28 Days Following the Study Intervention Dose | 28 days
Severity of Unsolicited NOCIs for 28 Days Following the Study Intervention Dose | 28 days
Geometric Mean Titer (GMT) at Day 0 of Serum Functional Antibody Against GI.1 Measured by Norovirus Blocking Antibody Assay (NBAA) | Day 0
GMT at Day 28 of Serum Functional Antibody Against GI.1 Measured by NBAA | Day 28
GMT at Day 0 of Serum Functional Antibody Against GII.4 Measured by NBAA | Day 0
GMT at Day 28 of Serum Functional Antibody Against GII.4 Measured by NBAA | Day 28
Geometric Mean Fold Rise (GMFR) from Day 0 to Day 28 of Serum Functional Antibody Against GI.1 Measured by NBAA | From Day 0 to Day 28
GMFR from Day 0 to Day 28 of Serum Functional Antibody Against GII.4 Measured by NBAA | From Day 0 to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Johnson County Clin Trials - JCCT, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No